CLINICAL TRIAL: NCT00347763
Title: Strategies for the Control of Blinding Trachoma: Effect of Fly Spray
Brief Title: Effect of Intensive Fly Control on Trachoma and Ocular Chlamydia Infection in Tanzania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Wellcome Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WellcomeTrust 059134
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2004-05

CONDITIONS: Trachoma
Keywords: trachoma; chlamydia; flies; permethrin
MeSH Terms: conditions — Trachoma; Chlamydia Infections | interventions — Permethrin

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- control (No Intervention): no active fly spray intervention
- intervention (Active Comparator): aerial spray of permethrin daily for two weeks and weekly as needed by assessment of fly density
  Interventions: Procedure: 10% permethrin in water applied as low volume spray

INTERVENTIONS:
Procedure: 10% permethrin in water applied as low volume spray
  Arms: intervention

SUMMARY:
The purpose of this community-based randomized trial was to determine, in trachoma hyper-endemic communities of Tanzania, the added value of intensive spraying to control flies on the fly population and on trachoma and ocular chlamydia infection at 6 months and one year after mass antibiotic treatment.

DETAILED DESCRIPTION:
Trachoma is the leading infectious cause of blindness in the world. The World Health Organization (WHO), recognizing the important public health impact of trachoma, has adopted a resolution to eliminate blinding trachoma by the year 2020 (3). In order to accomplish this ambitious goal, WHO recommends the use of "SAFE" strategy for countries implementing trachoma control programs. This multi-faceted approach includes Surgery for trichiasis cases, Antibiotics to treat the community pool of infection, Face washing to reduce transmission, and Environmental change.

The environmental change component currently rests largely on efforts to reduce the fly populations in these communities. A pilot study and clinical trial using intense insecticide spraying reduced both flies and trachoma in a trachoma hypo-endemic area of The Gambia. In The Gambia setting, flies appear to be an important vector for trachoma, but it is not clear that flies are equally important in areas with hyper-endemic trachoma, nor is it known if fly control adds value to the provision of mass antibiotic treatment for active trachoma as part of the SAFE strategy.

The purpose of this community-based randomized trial was to determine, in trachoma hyper-endemic communities of Tanzania, the added value of intensive spraying to control flies on the fly population and on trachoma and ocular C. trachomatis infection at 6 months and one year after mass antibiotic treatment. Neighborhoods with intensive spraying (Intervention) and neighborhoods with no spraying (control) all received mass antibiotic treatment with azithromycin immediately prior to the start of the study, enabling us to evaluate the additional impact of fly control on trachoma.

Kongwa district in central Tanzania has been shown to have a high prevalence of active trachoma, and was chosen as the site of this study. We randomized sixteen balozi to receive either mass treatment with azithromycin alone (control), or mass treatment plus an intensive fly spraying program (intervention). Pre-school aged children are the reservoirs of infection and disease within these communities. Therefore, within each balozi, all children aged less than eight served as sentinel markers for the status of trachoma at baseline, 6 months, and one year after baseline. In the eight intervention balozi, 119 children from 87 families were enrolled at baseline, and in the eight control balozi, 183 children from 145 families were enrolled.

The balozis were surveyed and an area surrounding the intervention balozis was targeted for insecticide spray. A solution of 10% permethrin in water was used with a Hudson and MicronAir sprayer machines, At the outset, spraying was carried out every two days for two weeks (attack phase) then once per week (maintenance phase) for the rest of the study.

Two sticky traps, fly paper strips were placed in each balozi to capture flies. The traps were changed every week, and the number of flies captured were counted. If the average number in the intervention balozis exceeded 25% of that in the control balozis, an attack phase, as described above, was reinstituted to keep the fly population low in the intervention group.

The primary outcome was the prevalence of trachoma in the pre-school aged children at 6 months and one year post mass antibiotic treatment.Outcomes are reported based on masked photographic gradings. Secondary outcome was ocular C. trachomatis infection, based on use of Amplicor C. trachomatis qualitative PCR assay.

comparison: Balozi randomized to receive intensive fly spray intervention,compared to Balozi with no fly spray intervention

ELIGIBILITY:
Inclusion Criteria:

* Balozi in Chiwe area
* Sentinel children: age less than 8 years

Exclusion Criteria:

* Balozi in Chiwe without geographic borders
* Sentinel children:age more than 8 years

Ages: 12 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350
Dates: Start 2000-06; Primary Completion 2002-09 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
clinical trachoma | 1 year
  clinical grading of conjunctival photographs for follicular trachoma

SECONDARY OUTCOMES:
ocular C. trachomatis infection | 6 months
  laboratory assessment of chlamydial DNA on ocular swab; measured as present or absent

CONTACTS AND LOCATIONS:
Overall Officials: Sheila West, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University/ Kongwa Trachoma Project, Baltimore, Maryland, United States

REFERENCES:
- [Result] West SK, Emerson PM, Mkocha H, McHiwa W, Munoz B, Bailey R, Mabey D. Intensive insecticide spraying for fly control after mass antibiotic treatment for trachoma in a hyperendemic setting: a randomised trial. Lancet. 2006 Aug 12;368(9535):596-600. doi: 10.1016/S0140-6736(06)69203-9. PMID 16905024